CLINICAL TRIAL: NCT03525730
Title: LRAs United as a Novel Anti-HIV Strategy (LUNA): a Randomized Controlled Trial.
Brief Title: LRAs United as a Novel Anti-HIV Strategy.
Acronym: LUNA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Casper Rokx, MD PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-002837-48
Record Dates: First submitted 2018-04-23; First posted 2018-05-16 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: HIV-1-infection
Keywords: HIV; Latency reversing agents; HDAC inhibitor; BAF inhibitor; HIV reservoir; HIV cure
MeSH Terms: interventions — Valproic Acid; Pyrimethamine

STUDY DESIGN:
Intervention Model Description: 6 week study, including 2 week intervention and 4 week post-treatment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Control (No Intervention): This group receives no intervention.
- Valproic acid (Experimental): This group receives valproic acid (enteric) for 14 days.
  Interventions: Drug: Valproic Acid
- Pyrimethamine (Experimental): This group receives pyrimethamine for 14 days.
  Interventions: Drug: Pyrimethamine
- Valproic acid and Pyrimethamine (Experimental): This group receives valproic acid and pyrimethamine for 14 days.
  Interventions: Drug: Valproic Acid; Drug: Pyrimethamine

INTERVENTIONS:
Drug: Valproic Acid — Valproic acid (enteric) 30mg/kg, divided over 2 doses per day, orally on day 1-14.
  Other Names: Depakine
  Arms: Valproic acid; Valproic acid and Pyrimethamine
Drug: Pyrimethamine — Pyrimethamine 200mg once daily (QD) orally on day 1 and 100mg on day 2-14.
  Other Names: Daraprim
  Arms: Pyrimethamine; Valproic acid and Pyrimethamine

SUMMARY:
A translational proof of concept study in humans on the primary research question whether novel anti-human immunodeficiency virus (HIV) latency strategies, including a BAF inhibitor and a histone deacetylase inhibitor, result in HIV reservoir reduction in HIV patients on antiretroviral therapy.

DETAILED DESCRIPTION:
The retrovirus HIV integrates as proviral DNA in the genome of cluster of differentiation (CD)4+ T cells. A subset form a reservoir of latently infected long-lived memory T-cells with nearly absent HIV-DNA transcription. This persistent latent HIV reservoir is the major obstacle for a cure. HIV latency is sustained by multiple host factors that restrict the viral promotor and expression of the viral genome. Latency reversing agents (LRA) can remove these restrictive components and mediate HIV latency reversal. LRA monotherapy with histone deacetylase inhibitors (HDACi) alone, including valproic acid, vorinostat, romidepsin, or panobinostat, reactivate HIV but seems insufficient to eliminate the reservoir in vivo. Our research group has identified the BAF complex as another repressive factor that maintains HIV latency. Pyrimethamine acts as an inhibitor of this BAF complex, is capable of reactivating HIV from latency at clinical tolerable concentrations, and acts synergistic with other LRA classes. This offers new opportunities for cure research. This is the first translational clinical study with BAF inhibitors and it assesses the potential synergism of 2 LRA with different modes of action on the reservoir in HIV patients.

Primary objective:

The longitudinal assessment of the effects of the BAF inhibitor pyrimethamine and of the HDACi valproic acid on the HIV reservoir in HIV patients on antiretroviral therapy.

Study design:

Open label 6 week randomized controlled intervention trial.

Study population:

Participants must be HIV infected, ≥18 years and on antiretroviral therapy with plasma HIV-RNA <50 copies/mL and CD4+ T cell count ≥200 cells/mm3 at enrollment. The HIV-RNA was ≥10.000 copies/mL before antiretroviral therapy initiation.

Intervention:

Participants are randomized to either of 4 arms and receive valproic acid, pyrimethamine, both for 2 weeks, or no intervention. Total study duration is 6 weeks and includes a 2 week treatment period and a 4 week post-treatment period.

Primary endpoint:

The change in HIV reactivation in the reservoir in vivo at treatment initiation and at the end of treatment, measured as the change in cell associated HIV-RNA. The change in reactivation is compared between the treatment arms.

Secondary endpoints:

See below.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected patients ≥18 years.
2. World Health Organization (WHO) performance status 0 or 1.
3. Confirmed HIV-1 infection by 4th generation ELISA, Western Blot or PCR.
4. Wild type HIV infection or polymorphisms associated with at highest low-level resistance to any class of ART according to Stanford HIV drug resistance database. Transmitted mutations and acquired mutations due to virological failure associated with resistance of at highest low-level resistance are allowed.
5. On cART.
6. Current plasma HIV-RNA <50 copies/mL for at least 365 days and measured on at least 2 occasions of which at least 1 must be obtained within 365 and 90 days prior to study entry.
7. Current CD4 T-cell count at study entry of ≥200 cells/mm3.
8. Pre-cART HIV-RNA ≥10.000 copies/mL.

Exclusion Criteria:

1. Previous virological failure, defined as either acquired resistance mutations (>low level resistance) on cART or HIV-RNA >1000 copies/mL on two consecutive measurements during cART.
2. Uncontrolled hepatitis B or C co-infection. For hepatitis B: patients should be vaccinated, or on pre-exposure prophylaxis through the use of lamivudine/emtricitabine or tenofovir in their combination ART. Otherwise, standard serological testing should be available within the last 365 days for homosexual HIV positive men. For non-homosexual HIV positive persons, there should be at least one negative hepatitis B test (either by serology or PCR). For homosexual HIV positive men, a negative hepatitis C immunoglobulin G, hepatitis C (HCV) antigen, blot or HCV-RNA PCR should be available within the previous 365 days. For non-homosexual HIV positive persons, there should be at least one negative hepatitis C test (either IgG, blot or PCR) available.
3. Prior exposure to any HDACi, BAFi or other known LRA.
4. Prior exposure to cytotoxic myeloablative chemotherapy for hematological malignancies during cART.
5. Concurrent exposure to strong interacting medication on glucuronidation.
6. Exposure within 90 days prior to study entry to immunomodulators, cytokines, systemic antifungals, dexamethasone, vitamin K antagonists, anti-epileptics, antipsychotics, carbapenems, mefloquine, colestyramine, Any documented opportunistic infection related to HIV in the last 90 days.
7. Inadequate blood counts, renal and hepatic function tests

   1. Haemoglobin <6.5 mmol/L (males) or <6.0 mmol/L (females), leucocytes <2.5 x109/L, absolute neutrophil count <1000 cells/mm3, thrombocytes <100 x109/L, international standardized ratio >1.6, activated partial thromboplastin time >40 seconds.
   2. Estimated glomerular filtration rate <50 mL/min (CKD-EPI),
   3. Alanine aminotransferase or total bilirubin >2.5x upper limit of normal.
   4. All laboratory values must be obtained within 42 days prior to the baseline visit.
8. Megaloblastic anemia due to folate deficiency.
9. Pancreatitis in last 6 months, or chronic pancreatitis.
10. Active malignancy during the past year with the exception of basal carcinoma of the skin, stage 0 cervical carcinoma, Kaposi Sarcoma treated with cART alone, or other indolent malignancies.
11. Females in the reproductive age cannot participate. Males cannot participate if they refuse to abstain from sex or condom use in serodiscordant sexual contact during the study, except if their sexual partner(s) use pre-exposure prophylaxis.
12. Patients with active substance abuse or registered allergies to the investigational medical products.
13. Last, any other condition (familial, psychological, sociological, geographical) which in the investigator's opinion poses an unacceptable risk or would hamper compliance with the study protocol and follow up schedule, will prohibit participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Cell associated HIV-RNA | 6 week
  The change in cell associated HIV-RNA between treatment initiation (week 0) and at the end of study (week 6). The change wil be compared between the study arms.

SECONDARY OUTCOMES:
Tat/rev induced limiting dilution assay (TILDA) | 6 week
  The change in TILDA between the groups between week 2 and week 0, between week 6 and week 2, and between week 6 and week 0 The change will be compared between the study arms.
Synergy | 6 week
  Potential synergism or additive effects of the administration of both drugs will be assessed by performing separate models including either both treatments or separate and subsequently investigating which model best predicts the outcome. the Bliss independence method to assess synergism will be performed. The combination therapy is considered synergistic if the difference and its 95% normal confidence interval (CI) were >0.
Cell associated HIV-RNA | 6 week
  The change in cell associated HIV-RNA between and within the groups between week 2 and week 0, between week 6 and week 2, and between week 6 and week 0.
Cell associated HIV-DNA | 6 week
  The change in cell associated HIV-DNA between and within the groups between week 2 and week 0, between week 6 and week 2, and between week 6 and week 0.
Plasma HIV-RNA | 6 week
  The change in plasma HIV-RNA between and within the groups between week 2 and week 0, between week 6 and week 2, and between week 6 and week 0.
Histone deacetylation | 6 week
  The change in the level of histone acetylation between and within the groups between week 0 and week 2, and between week 2 and week 6.
Expression of BAF subunits | 6 week
  The change in the level of expression between and within the groups between week 0 and week 2, and between week 2 and week 6.
Immunological functionality | 6 week
  The change of the functionality of innate immune cells, HIV specific CD4+ and CD8+ T cells and HIV specific B-cells between and within the groups between week 0 and week 2, and between week 2 and week 6.
Immunological cytotoxicity | 6 week
  The change of the cytotoxicity of innate immune cells, HIV specific CD4+ and CD8+ T cells and HIV specific B-cells between and within the groups between week 0 and week 2, and between week 2 and week 6.
Immunological phenotype | 6 week
  The change of the phenotype of innate immune cells, HIV specific CD4+ and CD8+ T cells and HIV specific B-cells between and within the groups between week 0 and week 2, and between week 2 and week 6.
Reservoir biomarkers | 6 week
  The correlations between clinical markers, markers of the viral reservoir (HIV-DNA, HIV-RNA), frequency and functionality of immune cells, cytokines, and level of acetylation/BAF expression with the change in reservoir (cell asociated-HIVRNA and TILDA) within and between the treatment arms
In vivo/ex vivo reservoir reactivation correlation | 6 week
  The correlation between ex vivo/in vitro (primary CD4 T cells, and cell line based) LRA efficacy, assessed using the size of the reservoir as measured by TILDA, HIV-DNA, HIV-RNA and level of acetylation/BAF expression after stimulation by pyrimethamine, valproic acid or both, and this will be correlated to these observed reservoir measurements outcomes in vivo at week 2 and week 6.
Incidence of Treatment-Emergent Adverse Events | 6 week
  The clinical and biochemical adverse events will be assessed by the Common Toxicity Criteria.
Plasma HIV-RNA | 6 week
  The proportion of subjects with plasma HIV-RNA >=20, >=50, >=200 at weeks 0, weeks 2 and week 6.
Pharmacokinetics of dolutegravir | 6 week
  Plasma concentrations Cmax dolutegravir will be measured using validated methods in patients receiving these medications. The pharmacokinetic profiles of the dolutegravir will be assessed in relation to the primary endpoint and use of valproic acid.
Pharmacokinetics of dolutegravir | 6 week
  Plasma concentrations Ctrough dolutegravir will be measured using validated methods in patients receiving these medications. The pharmacokinetic profiles of the dolutegravir will be assessed in relation to the primary endpoint and use of valproic acid.
Pharmacokinetics of valproic acid | 6 week
  Plasma concentrations Ctrough of valproic acid will be measured using validated methods in patients receiving these medications. The total and free (nonprotein-bound) plasma concentrations of valproic acid will be measured. The pharmacokinetic profiles of the investigational medical products will be assessed in relation to the primary endpoint.
Pharmacokinetics of valproic acid | 6 week
  Plasma concentrations Cmax of valproic acid will be measured using validated methods in patients receiving these medications. The total and free (nonprotein-bound) plasma concentrations of valproic acid will be measured. The pharmacokinetic profiles of the investigational medical products will be assessed in relation to the primary endpoint.
Pharmacokinetics of pyrimethamine | 6 week
  Plasma concentrations Cmax of pyrimethamine will be measured using validated methods in patients receiving this medication. The pharmacokinetic profiles of the investigational medical products will be assessed in relation to the primary endpoint.
Pharmacokinetics of pyrimethamine | 6 week
  Plasma concentrations Ctrough of pyrimethamine will be measured using validated methods in patients receiving this medication. The pharmacokinetic profiles of the investigational medical products will be assessed in relation to the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Casper Rokx, MD PhD, Principal Investigator — Erasmus Medical Center; Tokameh Mahmoudi, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
No definitive decision on this yet. This will also depend on confidentiality.

REFERENCES:
- [Derived] Bollen PDJ, Prins HAB, Colbers A, Velthoven-Graafland K, Rijnders BJA, de Vries-Sluijs TEMS, van Nood E, Nouwen J, Bax H, de Mendonca Melo M, Verbon A, Burger DM, Rokx C. The dolutegravir/valproic acid drug-drug interaction is primarily based on protein displacement. J Antimicrob Chemother. 2021 Apr 13;76(5):1273-1276. doi: 10.1093/jac/dkab021. PMID 33544819